CLINICAL TRIAL: NCT04554940
Title: A Randomized, Controlled, Open-label Clinical Trial With an Open-label Extension to Investigate the Safety of Vosoritide in Infants and Young Children With Achondroplasia at Risk of Requiring Cervicomedullary Decompression Surgery
Brief Title: A Clinical Trial to Evaluate Safety of Vosoritide in At-risk Infants With Achondroplasia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 111-209
Record Dates: First submitted 2020-09-14; First posted 2020-09-18 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Achondroplasia
Keywords: Dwarfism; Bone Diseases; Bone Diseases, Developmental ACH; Natriuretic Peptide, C-Type; Musculoskeletal Diseases
MeSH Terms: conditions — Achondroplasia; Dwarfism; Bone Diseases; Musculoskeletal Diseases | interventions — vosoritide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Vosoritide + Standard of Care (Experimental): Standard of Care treatment for cervicomedullary compression and once daily subcutaneous injection of recommended dose of vosoritide based on weight-band dosing.
  Interventions: Biological: vosoritide
- Standard of Care Alone (No Intervention): Institutional standard of care monitoring and treatment for cervicomedullary compression

INTERVENTIONS:
Biological: vosoritide — Subcutaneous injection of recommended dose of BMN 111 based on weight-band dosing once daily.
  Arms: Vosoritide + Standard of Care

SUMMARY:
Study 111-209 is a Phase 2 randomized, open-label clinical trial of BMN 111 in infants and young children with a diagnosis of Achondroplasia at a heightened risk of requiring cervicomedullary decompression surgery

ELIGIBILITY:
Inclusion Criteria:

* Parent(s) or guardian(s) willing and able to provide signed informed consent after the nature of the study has been explained and prior to performance of any research related procedure.
* Have ACH, documented by genetic testing.
* Are willing and able to perform all study procedures as physically possible.
* Age 0 to ≤ 12 months, at study entry (Day 1). Given that any potential impact of vosoritide therapy on the foramen magnum is dependent on treating as early as possible and as long as possible while the synchondroses at the base of the skull are still open. For subjects > 6 months of age at enrollment, a discussion between the investigator and the Medical Monitor should occur with the goal of limiting the number of subjects in the range of > 6 months to ≤ 12 months of age.
* Parent(s) or caregiver(s) are willing to administer daily injections to the subject and complete the required training.
* Have evidence of CMC that "may" require surgical intervention

Exclusion Criteria:

* Have hypochondroplasia or short-stature condition other than achondroplasia (eg, trisomy 21, pseudoachondroplasia, etc).
* Have CMC that either does not require surgical intervention (for example foramen magnum narrowing with preservation of the cerebrospinal fluid space) or does require immediate surgical intervention .
* Have any of the following: Untreated congenital hypothyroidism or maternal history of hyperthyroidism, Insulin-requiring neonatal diabetes mellitus, Autoimmune inflammatory disease, Inflammatory bowel disease, Autonomic neuropathy.
* Have a history of any of the following:Renal insufficiency, Chronic anemia,Baseline systolic blood pressure below age and gender specified normal range or recurrent symptomatic hypotension (defined as episodes of low blood pressure generally accompanied by symptoms eg, pallor, cyanosis, irritability, poor feeding) and Cardiac or vascular disease.
* Have a clinically significant finding or arrhythmia that indicates abnormal cardiac function or conduction or QTc-F ≥ 450 msec on screening ECG.
* Have been treated with growth hormone, insulin-like growth factor 1, or anabolic steroids in the 6 months prior to Screening, or long-term treatment (> 3 months) at any time.
* Have ever had prior cervicomedullary decompression surgery.
* Have had a fracture of the long bones or spine within 6 months prior to Screening.

Ages: 0 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Through Week 260

SECONDARY OUTCOMES:
Evaluate the effect of Vosoritide on total foramen magnum volume (in cm3) by MRI volumetric measurement software | Through Week 260

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — BioMarin Pharmaceutical
Locations (3):
- Murdoch Children's Research Institute, Parkville, Victoria, Australia
- United Kingdom (2):
  - Guy's and St. Thomas NHS Foundation Trust Evelina Children's Hospital, London
  - Sheffield Children's NHS Foundation Trust, Sheffield

REFERENCES:
- [Derived] Savarirayan R, Irving M, Maixner W, Thompson D, Offiah AC, Connolly DJ, Raghavan A, Powell J, Kronhardt M, Jeha G, Ghani S, Fisheleva E, Day JR. Rationale, design, and methods of a randomized, controlled, open-label clinical trial with open-label extension to investigate the safety of vosoritide in infants, and young children with achondroplasia at risk of requiring cervicomedullary decompression surgery. Sci Prog. 2021 Jan-Mar;104(1):368504211003782. doi: 10.1177/00368504211003782. PMID 33761804